CLINICAL TRIAL: NCT03404427
Title: Effects of Sleep Privation on Sensorimotor Integration of the Upper Limb During a Manual Endurance Test in Healthy Volunteers-Physiological Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HANDY-SLEEP
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Sleep Deprivation; Healthy Volunteers; Skeletal Muscle
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: To compare the motor endurance of healthy subjects after a normal sleep night and after a sleepless night.
Who Masked: Outcomes Assessor
Masking Description: When analyzing the results (endurance, magnitude of the premotor potential), the outcomes assessor will not know if it is a normal night or a sleepless night
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal sleep night (Sham Comparator): The first endurance test is the endurance motor control test after a normal sleep night.
  Interventions: Behavioral: Normal sleep night
- Sleepless night (Experimental): The first endurance test is the endurance motor test after a sleepless night.
  Interventions: Behavioral: Sleepless night

INTERVENTIONS:
Behavioral: Normal sleep night — Usual hours of sleep
  Arms: Normal sleep night
Behavioral: Sleepless night — Total sleep deprivation the first night
  Arms: Sleepless night

SUMMARY:
The investigator showed that a night of sleep deprivation halved the duration of an inspiratory endurance test and that this loss of endurance could be secondary to a lack of activation of the pre-motor cortex. However, the inspiratory endurance test is associated with a feeling of dyspnea that could lead to premature arrest, and the inspiratory drive is complex, both automatic and voluntary. The investigator can reproduce this results on a simpler drive.

During the execution of an exercise involving repeated contractions of the hand it is possible to record the activation of the pre-motor cortex corresponding to the phase of preparation of the movement. The amplitude of these premotor potentials is proportional to the developed motive force.

The purpose of this study is to assess the impact of sleep deprivation on the muscular endurance of non-dominant in healthy subjects.

Hypothesis: Sleep deprivation causes a decrease in manual motor endurance by decreasing cortical pre-motor control.

Main objective: To compare the motor endurance of healthy subjects after a night's sleep and after a sleepless night.

Secondary objective: To compare the amplitude of premature cortical control at the beginning of the endurance test after a night's sleep and after a sleepless night.

ELIGIBILITY:
Inclusion Criteria:

* adult male volunteers;
* 25 to 45 years old
* regularly sleeping more than 6 hours per night;
* no excessive consumers of coffee (<3 espressos / day);
* absence of muscular or neurological pathology ;
* with a BMI> 18 and <25 kg / m²;
* Horne and Ostberg score> 31 and <69 ;

Exclusion Criteria:

* female sex
* history of neuromuscular disease ;
* implanted metallic or electronic equipment (vascular stent, ocular implant, pacemaker ...)
* history of epilepsy, or discomfort after sleep deprivation ;
* poor sleepers (PSQI> 5);
* exercising an activity in staggered hours;
* regularly performing more than 2 nights without sleep per month;
* taking drugs interfering with sleep (antidepressants, benzodiazepines ...);
* having crossed 4 time zones in the previous 4 weeks.
* current participation in another clinical research study;

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Test duration | 1 hour.
  Time, in minutes, measured between the beginning of the endurance test and the end of the test, defined by the volunteer's inability to maintain a force of at least 30% of the maximum strength for 5 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Drouot, Principal Investigator — Poitiers University Hospital
Locations (1):
- Centre Hospitalier de Poitiers, Poitiers, Vienne, France

REFERENCES:
- [Derived] Rault CCS, Heraud Q, Ansquer S, Ragot S, Kostencovska A, Thille AW, Stancu A, Saulnier PJ, Drouot X. Sleep Deprivation in Healthy Males Increases Muscle Afferents, Impairing Motor Preparation and Reducing Endurance. J Clin Neurophysiol. 2024 Nov 27;42(5):457-465. doi: 10.1097/WNP.0000000000001134. PMID 39593197